CLINICAL TRIAL: NCT00582283
Title: NM404 as an Imaging Agent in Patients With Non-small Cell Lung Cancer (NSCLC)
Brief Title: NM404 as an Imaging Agent in Patients With NSCLC
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Cellectar Biosciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CO02505; R21CA092412 (NIH); 124I-CLR1404 (Other Grant/Funding Number: Novelos Therapeutics)
Record Dates: First submitted 2007-12-19; First posted 2007-12-28 (Estimated); Last update posted 2019-05-22 (Actual); Status verified 2019-05

CONDITIONS: Non Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Diagnostic: iodine I-124 NM404 CT/PET scan (Other): Patients undergo iodine I-124 NM404 CT/PET scan at 1-2, 4-6, 24, and 48 hours and at 5-10 days.
  Interventions: Drug: I124-NM404

INTERVENTIONS:
Drug: I124-NM404 — I-124-NM404

SUMMARY:
This study seeks to determine imaging characteristics of radiolabelled 131-I-NM404 in ten patients with cancer, including calculations of PKs, radiation dosimetry, biodistribution, and optimal imaging times (part 1 - complete).

In addition, specific tumor accumulation and metabolic fate of 131-I-NM404 will be determined in NSCLC tumors collected in 5 patients (part 2 - complete). Lastly, the study will collect preliminary data on imaging NSCLC tumors in up to 12 patients with evaluable disease (part 3 - ongoing).

ELIGIBILITY:
Inclusion Criteria: Part 3

* Histologically or cytologically documented NSCLC with measurable of disease
* Disease is evaluable by CT scan
* At least 18 years old. Women cannot be pregnant or breastfeeding
* Karnofsky score >/= to 60
* Adequate renal/hepatic function
* Adequate blood cell count levels

Exclusion Criteria:

* Concomitant infection
* Other active cancers

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2004-01-14 (Actual); Primary Completion 2014-08-01 (Actual); Study Completion 2014-08-01 (Actual)

PRIMARY OUTCOMES:
Qualitative Image Analysis of NSCLC tumors with 124I-NM404 imaging agent | 5 days
  The objective of this protocol is to obtain preliminary data on imaging NSCLC tumors. Images with 124I-NM404 will be evaluated by a nuclear medicine consultant, who will be blind to the participants' clinical findings and other radiographic images. The nuclear medicine consultant will independently record his findings, and then compare his results with those obtained by conventional FDG-PET imaging that was done at baseline as part of this study. This comparison will be only qualitative.

SECONDARY OUTCOMES:
Semi-quantitative lesion scoring to evaluate Tumor biodistribution | up to 7 days
  Images will be evaluated by physician who will be blinded to the participants' clinical or CT findings. The physician will score scans at the various time points for intensity of tumor uptake. A typical 0-3 scale will be used: 0 = no perceptible uptake, 1+ = uptake barely perceptible above background, 2+ = uptake clearly distinguishable above background, 3+ = intense uptake, much greater than surrounding normal structures (2+ and 3+ are considered abnormal or positive for lesion identification; 0 and 1+ are considered normal or negative for lesion identification).

CONTACTS AND LOCATIONS:
Overall Officials: Anne M Traynor, MD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin Carbone Comprehensive Cancer Center, Madison, Wisconsin, United States